CLINICAL TRIAL: NCT04477434
Title: Observatoire National d'ElectroConvulsivoThérapie (ECT)
Brief Title: French Observatory of ElectroConvulsive Therapy (ECT)
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Other Study IDs: 2035305v1
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the 30s, ECT has been a psychiatric treatment mainly used for drug-resistant depressive illnesses. Clinical studies have shown its therapeutic efficiency compared to standard treatments also in other psychiatric illnesses. Although efficient, ECTs also induce side effects. In France, there is currently no consensus on providing the suitest medical care. It is therefore important to review our nowadays health care models in order to maintain and improve the recommendations of the French National Agency for Accreditation and Evaluation in Health, the last of which date from 1997! Within this context, this project has the dual objective of (1) identifying ECT medical procedure in France and (2) developing research to evaluate and to improve the effectiveness of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively referred for ECT.

Exclusion Criteria:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving ECT as part of their medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ECT efficiency on patients | 2018-2022

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - CHU d'Angers : Site Larrey, Angers
  - Clinique Mirambeau, Anglet
  - CHS de Montfavet, Avignon
  - CH Cote Basque, Bayonne
  - Fondation bon sauveur, Bégard
  - Centre de crise Esquirol, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CH La Chartreuse, Dijon
  - Clinique du domaine de Vontes, Esvres-sur-Indre
  - Clinique de Pen-An-Dalar, Guipavas
  - CUMP Océan Indien, La Réunion
  - CH Marius Lacroix, La Rochelle
  - Césame, Les Ponts-de-Cé
  - CH de Mayenne, Mayenne
  - CHR Metz-Thionville, Metz
  - CH psy de la drôme Vivarais, Monteléger
  - CHS la Colombiere, Montpellier
  - CH Saint Roch, Nice
  - CH Sainte Anne, Paris
  - CH Henri Laborit, Poitiers
  - CHI Redon-Carentoir, Redon
  - CH Guillaume Regnier, Rennes
  - CH du Rouvray, Rouen
  - Epsm du Morbihan, Saint-Avé
  - Clinique Villa du Parc, Saujon
  - CH Civil 1, Strasbourg
  - CH Nord Deux Sèvres, Thouars
  - CHITS CH Sainte Musse, Toulon
  - CH Purpan, Toulouse
  - CPU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided